CLINICAL TRIAL: NCT03360006
Title: A Phase 1 Study Evaluating the Safety and Pharmacokinetics of ABBV-744 in Subjects With Relapsed/Refractory Acute Myeloid Leukemia (AML)
Brief Title: A Study Evaluating the Safety and Pharmacokinetics of ABBV-744 in Participants With Relapsed/Refractory Acute Myeloid Leukemia (AML) Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic Reasons
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M16-415
Record Dates: First submitted 2017-11-28; First posted 2017-12-02 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: Acute Myeloid Leukemia (AML); Relapsed/refractory acute myeloid leukemia; Dose-limiting toxicity; Recommended phase two dose; Pharmacokinetics
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — ABBV-744

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ABBV-744 Dose Escalation (Experimental): ABBV-744 will be administered at escalating dose levels until the maximum tolerated dose is reached and a recommended Phase 2 dose is determined.
  Interventions: Drug: ABBV-744
- ABBV-744 Dose Expansion (Experimental): ABBV-744 will be administered at the recommended Phase 2 dose determined during the Dose Escalation phase.
  Interventions: Drug: ABBV-744

INTERVENTIONS:
Drug: ABBV-744 — Tablet, oral

SUMMARY:
This is an open-label, Phase 1, dose-escalation (Segment 1) and expansion (Segment 2) study to determine the maximum tolerated dose (MTD) and/or the recommended phase two dose (RPTD), and to assess the safety, preliminary efficacy, and pharmacokinetic (PK) profile of ABBV-744 in participants with relapsed/refractory Acute Myeloid Leukemia (AML).

ELIGIBILITY:
Inclusion Criteria:

* Participant must have AML not amenable to curative therapy, refractory to standard of care therapy or for which standard of care therapy does not exist. Participants who are candidates for stem cell transplantation must have been offered this therapeutic option.
* Must consent to provide biomarker analyses as described in the protocol.
* Must have an Eastern Cooperative Oncology Group (ECOG) Performance status of:

  * Dose Escalation (Segment 1): 0 - 1
  * Dose Expansion (Segment 2): 0 - 2
* Dose Escalation: Must have a serum albumin during Screening of >= 3.0 g/dL.
* Participant has adequate bone marrow, renal and hepatic function.

Exclusion Criteria:

* Participant with known active Central Nervous System (CNS) disease.
* Participant has received anti-cancer traditional medicine or anti-cancer herbal remedies within 14 days prior to ABBV-744 dosing. Saw palmetto is considered anti-cancer herbal remedy. Participant has received anti-cancer therapy within a period of 14 days or 5 half-lives (whichever is longer; except for immunotherapy where a period of 21 days will be acceptable) prior to Study Day 1. Except for hydroxyurea which will be allowed during screening and treatment for controlling leukocytosis.
* Participant has been previously treated with a Bromodomain and Extra-Terminal (BET) inhibitor
* Participant has unresolved clinically significant toxicities from most recent prior anti-cancer therapy, defined as any Common Terminology Criteria for Adverse Events (CTCAE v 4.03) grade 2 or higher clinically significant toxicity (excluding alopecia).
* Participant has received the following within 7 days prior to the first dose of study drug: corticosteroid therapy, CYP3A inhibitors, CYP3A inducers.
* Participant consumed grapefruit or grapefruit products within 3 days prior to the first dose of study drug.
* Participant had major surgery within 28 days prior to Study Day 1.
* Participant is unable to swallow or absorb oral tablets.
* Participant has known infection with hepatitis B or hepatitis C.
* Participant has active peptic ulcer disease or other hemorrhagic esophagitis/gastritis, enteritis, colitis.
* Participant has symptoms of gross hematuria or gross hemoptysis
* Has electrocardiogram with a QT interval corrected for heart rate using Fridericia's formula (QTcF) > 470 msec or ECG with second degree type 2 or third degree atrioventricular block.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2020-12-19 (Actual); Study Completion 2020-12-19 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of ABBV-744 | Through Cycle 2 ( each cycle is 28 days)
  Cmax of ABBV-744.
Time to Cmax (Tmax) of ABBV-744 | Through Cycle 2 ( each cycle is 28 days)
  Tmax of ABBV-744.
Area under the plasma concentration-time curve (AUC) from time 0 to the time of the last measurable concentration (AUCt) of ABBV-744 | Through Cycle 2 ( each cycle is 28 days)
  Area under the plasma concentration-time curve (AUC) from time 0 to the time of the last measurable concentration (AUCt) of ABBV-744.
Terminal Phase Elimination Rate Constant (β) of ABBV-744 | Through Cycle 2 ( each cycle is 28 days)
  Terminal Phase Elimination Rate Constant (β) of ABBV-744.
Area under the plasma concentration-time curve (AUC) from time 0 to infinity (AUCinf) of ABBV-744 | Through Cycle 2 ( each cycle is 28 days)
  Area under the plasma concentration-time curve (AUC) from time 0 to infinity (AUCinf) of ABBV-744.
Dose-limiting toxicity (DLT) of ABBV-744 | Up to 28 days after first dose of study drug
  DLT events are defined as clinically significant adverse events or abnormal laboratory values assessed as unrelated to disease progression, underlying disease, intercurrent illness, or concomitant medications and occurring during the first 4 weeks after administration of the first dose and that meets additional criteria as described in the protocol.
Maximum Tolerated Dose (MTD) for ABBV-744 | Up to 28 days after first dose of study drug
  The MTD is defined as the highest dose for which the estimated posterior mean DLT rate is <= 33% and excessive toxicity probability is limited to maximum of 25% during the first 28 days.
Recommended Phase 2 Dose (RPTD) for ABBV-744 | Up to 28 days after first dose of study drug
  RPTD will be determined from a review available safety, pharmacokinetic, and efficacy data during the dose escalation phase (Segment 1) of the study.

SECONDARY OUTCOMES:
Composite complete remission (CRc) | Up to 2 years
  Percentage of participants who achieve composite complete remission (CRc), comprised of complete remission (CR) + CR with incomplete blood count recovery (CRi) is based on the International Working Group (IWG) criteria and European Leukemia Net criteria.
Complete Remission (CR) + CR with partial hematologic recovery (CRh) | Up to 2 years
  Percentage of participants who achieve CR + CR with partial hematologic recovery (CRh) is based on the International Working Group (IWG) criteria and European Leukemia Net criteria.
Objective Response Rate (ORR) | Up to 2 years
  Percentage of participants who achieve ORR [composite complete remission (CRc) + Partial remission (PR)] is based on the International Working Group (IWG) criteria (CRc, PR) and European Leukemia Net criteria.
Duration of Response (DOR) | Up to 2 years
  DOR is defined as the number of days from the date of first response to the first occurrence of progression or death from any cause, whichever occurs first.
Event-free survival (EFS) | Up to 2 years
  Percentage of participants who achieve EFS, where EFS is defined as the date of first dose of study drug to the date of primary refractory disease, relapse from CR or CRi, or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (7):
- United States (7):
  - UC Irvine /ID# 160789, Orange, California
  - University of California, Davis Comprehensive Cancer Center /ID# 202729, Sacramento, California
  - Northwestern /ID# 171098, Chicago, Illinois
  - University of Chicago DCAM /ID# 160702, Chicago, Illinois
  - Cleveland Clinic Main Campus /ID# 160756, Cleveland, Ohio
  - University of Texas MD Anderson Cancer Center /ID# 160701, Houston, Texas
  - Swedish-Center for Blood Disor /ID# 166487, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Crymes A, Evans MG, Jeyakumar D, Lou JJ, Zhao X, Rezk SA. Acute Myeloid Leukemia (AML) With T-Cell Differentiation Arising From Chronic Myelomonocytic Leukemia (CMML). Case Rep Hematol. 2024 Dec 14;2024:5584297. doi: 10.1155/crh/5584297. eCollection 2024. PMID 39734743
- [Derived] Zhang L, Cai T, Lin X, Huang X, Bui MH, Plotnik JP, Bellin RJ, Faivre EJ, Kuruvilla VM, Lam LT, Lu X, Zha Z, Feng W, Hessler P, Uziel T, Zhang Q, Cavazos A, Han L, Ferguson DC, Mehta G, Shanmugavelandy SS, Magoc TJ, Rowe J, Goodwin NC, Dorritie KA, Boyiadzis M, Albert DH, McDaniel KF, Kati WM, Konopleva M, Shen Y. Selective Inhibition of the Second Bromodomain of BET Family Proteins Results in Robust Antitumor Activity in Preclinical Models of Acute Myeloid Leukemia. Mol Cancer Ther. 2021 Oct;20(10):1809-1819. doi: 10.1158/1535-7163.MCT-21-0029. Epub 2021 Jul 12. PMID 34253595